CLINICAL TRIAL: NCT00616759
Title: The Effect on Cognition of Terminating ECT Induced Seizures With Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56164
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Major Depression
Keywords: Depression; Electroconvulsive therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Electroconvulsive Therapy; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ECT as usual
  Interventions: Procedure: electroconvulsive therapy
- 2 (Experimental): ECT-induced seizures terminated with propofol
  Interventions: Procedure: electroconvulsive therapy plus propofol; Drug: propofol

INTERVENTIONS:
Procedure: electroconvulsive therapy — electroconvulsive therapy as usual
  Arms: 1
Procedure: electroconvulsive therapy plus propofol — electroconvulsive therapy identical to the comparator group except that propofol 0.5 mg/kg is given intravenously 15 seconds after the electrical stimulation at each treatment in order to terminate the ECT-induced seizure
  Other Names: Diprivan
  Arms: 2
Drug: propofol — Propofol 0.5 mg/kg intravenously given 15 seconds following electrical stimulation
  Arms: 2

SUMMARY:
Participating subjects are those who are referred for electroconvulsive therapy (ECT) for severe depression who have agreed to the protocol. The control group receives ECT as usual. The other group receives propofol to terminate the ECT-induced seizure timed so that the seizure lasts at least 25 seconds. Extensive neuropsychological testing is being done on both groups before beginning ECT and within 48 hours after the 6th treatment. Multiple markers of the rapidity of recovery from anesthesia are being obtained from all subjects for 6 ECTs.

DETAILED DESCRIPTION:
ECT Administration All patients will receive ECT administered using a Thymatron-System IV (Somatics, LLC , Lake Bluff, IL) ECT device, the same device used for our usual ECT. All patients will be monitored with continuous electrocardiogram (EKG) monitoring, pulse oximetry, and regular blood pressure readings from an automatic inflatable cuff on one arm. Seizure threshold will be determined at the first treatment. The subsequent treatment will be administered at 1.5 times the seizure threshold. Stimulus dose will be increased as necessary to produce a seizure of at least 20 seconds observed duration of motor activity. All patients whose seizure duration is less than 20 seconds of motor activity will be re-stimulated at the same treatment session at a 50% increase in stimulus intensity unless this occurred at the maximum stimulus charge available. All monitoring described and the titration process is part of our normal ECT routine. Electrode placement will be bilateral for all patients which is the predominate placement used for our usual patients. Patients in the standard group will receive ECT as described elsewhere (Abrams, 2001). Patients in the experimental group will receive ECT as the other group. However, approximately 15 seconds after stimulus delivery they will receive a 1 mg/kg dose of propofol intravenously in order to terminate brain seizure activity reliably, whether evident on surface EEG or not. In view of 30-60 second circulation time this will limit seizure duration to 45-75 sec, and generally to the same duration at each session because the circulation time is an individual characteristic.

Routine anesthetic agents will include hyperventilation with 100% oxygen by mask, and initial dosages of succinylcholine 1 mg/kg IV, and etomidate 0.2 mg/kg IV, adjusted as needed over the treatment course. Atropine 0.4-1.0 mg will also be given intravenously before the anesthetic agent. Blood pressure and pulse will be assessed prior to treatment and 1 minute, 3 minutes, and 5 minutes following the ECT stimulus and periodically thereafter. All patients will receive at least 6 index ECT. Those needing additional treatment will receive standard ECT. Propofol and etomidate are used for our normal ECT treatments as well as atropine and succinylcholine. Blood pressure monitoring is also a part of routine ECT.

Electroencephalogram (EEG) Recording and Computer EEG Analysis Four channels of EEG data will be recorded using bilateral frontal-mastoid and bilateral frontal-occipital electrodes. Frontal and mastoid recording electrodes used will be EEG/EMG/ECG Adherent Recording Electrodes. (Somatics, LLC.) Occipital electrodes used will be Grass 10mm gold electrode. Preparation of the occipital area may include using Lemon Prep Skin Prep (Mavidon Medical LP-0019), Elefix conductive paste (Niho Kohden America, Inc.). Nu Prep Cover Roll stretch (BSN Medical) will be cut to facilitate the covering of electrodes. Analysis of some parameters of each seizure will be done with software provided by the manufacturer of the Thymatron system IV. Our standard ECT includes 2 channels of EEG recording using bilateral fronto-mastoid electrode placement using Adherent Recording Electrodes (Somatics, LLC) with computer analysis of channel 1.

Cognitive Assessment Cognition will be assessed using neuropsychological battery subtests which measure difficulties of retention of newly learned material (anterograde amnesia) and past events (retrograde amnesia) such as the California Verbal Learning Test (CVLT)(subtests: recognition tests A & B and long delay free recall). Wechsler Memory Scale (WMS III)(subtests: Mental Control, Logical Memory recognition, Memory Span), Trail Making A & B, Rey Auditory Verbal learning Test, and Rey Osterrieth Complex Figure Test (copy, recall and recognition trials). In addition, Hamilton Rating Scale of Depression, Clinical Global Improvement (CGI), Modified Mini Mental Status (3MSE), Autobiographical memory interview, Beck Depression Index (BDI) will be performed.

Emergence from anesthesia will be determined by measuring post-treatment reorientation time such as time to awaken, name recall, orientation to location, date and day of the week, with the time beginning at the end of stimulus application. Following awakening, patients will be asked at 1-min intervals to open their eyes and to squeeze the investigator's hand. The time from stimulation as well as the time from when the patients open their eyes to performance of the appropriate response to both commands will be noted. The same procedure will be used to identify place and date at 1-min intervals until the correct answer is given for each question. As soon as orientation occurs, we will administer a series of tests to evaluate recovery of psychomotor function, including the Trieger test (volunteers are asked to connect a series of dots), P-deletion test (volunteers are asked to select all letters "p" in a text of random letters during 180 s), and the Digit Symbol Substitution test (volunteers are asked to match numbers and symbols during 90 s) 15, 30, 45, 60, 75, and 90 min after cessation of anesthesia. These tests have been used previously to study recovery from anesthesia. At the same times patients will be asked to evaluate their "sense of clear-headedness," and "sense of energy". All assessments will be carried out by a blind investigator to the group membership of the patient. Our standard ECT utilizes the Mini Mental Status Examination before every third ECT to measure cognitive change. Cognitive testing emerging from anesthesia is not routinely done.

All subjects will receive six individual treatment sessions given 3 days per week. Investigators will be aware of the treatment parameters; however, independent raters will be blinded as to which treatment was administered.

Prior to the experimental treatment sessions, all subjects will participate in several preliminary meetings with the MD investigator and the psychologist. Each session will be used to facilitate the psychiatric screening, lab tests, psychological and neuropsychological tests in order to establish a baseline of memory functioning.

The experimental treatment sessions themselves will be supervised and facilitated by the MD investigator following the guidelines previously developed for this experimental procedure. Except for the administration of propofol or no drug at all following the administration of ECT, the treatment protocols will be exactly the same for each treatment group.

* All treatment sessions will begin will occur between 7:00 am and 12:00 pm and take place in the Loma Linda University Medical Center-Outpatient Surgery Center.
* Patients are instructed to not have anything to eat or drink (NPO) after midnight the night before ECT. They may take their morning blood pressure medications with a few sips of water.
* An intravenous (IV) line will be established. EEG Monitoring electrodes, O2 saturation monitor, and foot blood pressure cuff will be put in place. Atropine 0.4-1.0 mg IV will be administered first, then etomidate 0.2 mg/kg IV. Succinylcholine 1.0mg/kg IV will be given as soon as the patient falls asleep. Sleep will be measured by the inability to arouse the patient and the loss of the lash reflex. Other medications may be used to control blood pressure, nausea, etc.
* Patient will be masked with 100% O2 and hyperventilated
* Approximately ninety seconds after the infusion of succinylcholine, the impedance will be checked using the Thymatron and then the stimulus is given.
* During the first ECT session a titration procedure will be done in order to determine the lowest dose of electrical energy that will produce a seizure (seizure threshold).
* The second ECT is set at 50% above the seizure threshold.
* Subsequent stimulus settings are set to keep the seizure duration above 25 seconds at absolute minimum.
* Propofol 0.5-1.0 mg/kg will be administered IV to patients in the experimental group when the seizure duration reaches 15 seconds as measured by the EEG monitor at all of the first six ECTs, including at the session during which titration is done, and at the seventh ECT in the control group.
* Anesthesiologist will continue to mask the patient until the patient is able to adequately breathe on their own.
* Patient will be taken to the recovery area and monitored with O2 in place until stable.
* Time to awaken, time to name recall, place recall, and date recall will be assessed after each treatment by a rater who is blind to the treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth edition, Text Revision (DSM-IV-TR) criteria for major depression, single episode or recurrent
* Subjects must be over the age of 45 years
* Subjects must be willing to receive at least six treatments of ECT, along with pre ECT lab screening and pre and post psychological and neuropsychological tests
* The ability to read, speak and comprehend English and have the ability to complete the forms in writing
* Must be able to give consent for treatment
* Shorter acting benzodiazepines (aplrazolam, lorazepam) will be allowed on a prn basis but excluded 12 hours before each ECT session

Exclusion Criteria:

* Subjects who have a history of schizophrenia, bipolar affective disorder, delusional disorder, paranoid disorder, or schizoaffective disorder, or who are exhibiting psychotic symptoms [except mood congruent depressive delusions].
* Subjects who have a substance abuse/dependence disorder not in full remission
* Patients with significant medical problems that may increase risk or require unusual concomitant treatment
* Patients with significant neurological problems including seizure disorder
* Patients with a hearing or visual impairment that would interfere with the research process
* Patients with moderate to severe dementia. Any patient scoring less than 25 on the MMSE will have a Mattis Dementia Rating Scale-2 (DRS-2) test for dementia administered.
* Patients known to be intolerant of propofol, etomidate, or succinylcholine, or for whom these anesthetic medications are not appropriate
* Patients taking anticonvulsant medications such as Tegretol, Depakote, Klonopin, etc.
* Patients on an involuntary admission status
* Patients unable to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03-24 (Actual); Study Completion 2010-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L Warnell, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Result] Warnell RL, Swartz CM, Thomson A. Propofol interruption of ECT seizure to reduce side-effects: a pilot study. Psychiatry Res. 2010 Jan 30;175(1-2):184-5. doi: 10.1016/j.psychres.2009.08.019. Epub 2009 Nov 5. PMID 19892408

RESULTS

PARTICIPANT FLOW:
Groups:
- Series of 6 ECTs Performed With Standard Technique: Electroconvulsive Therapy (ECT) as usual
- 6 ECTs Where Seizure Was Shortened by Propofol: ECT-induced seizures terminated with propofol
Period: Overall Study
Arm/Group | Series of 6 ECTs Performed With Standard Technique | 6 ECTs Where Seizure Was Shortened by Propofol
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: PI left institution without completing results. Multiple attempts have been made to contact PI without success. No data available to submit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Series of 6 ECTs Performed With Standard Technique | 6 ECTs Where Seizure Was Shortened by Propofol | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Wechsler Memory Scale-III (WMS-III) Auditory Delayed Index
Description: WMS-III Auditory Delayed Index is a measure of memory functioning. The results given are the post-ECT testing results. A smaller number indicates less memory disturbance on this scale. The range of scores is between 0-140 with higher scores indicating better memory function.
Time Frame: Pre-tesing within 36 hours before first ECT; Post-testing within 36 hours of 6th ECT.
Population: PI left institution without completing results. Multiple attempts to contact PI have been unsuccessful. No data available to submit.
Arm/Group | Series of 6 ECTs Performed With Standard Technique | 6 ECTs Where Seizure Was Shortened by Propofol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: PI left institution without completing results. Multiple attempts to contact PI have been unsuccessful. No available data to submit.
Arm/Group | Series of 6 ECTs Performed With Standard Technique | 6 ECTs Where Seizure Was Shortened by Propofol
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No